CLINICAL TRIAL: NCT04237129
Title: A Glucose Clamp Trial Investigating The Biosimilarity of Gan & Lee Insulin Aspart Injection (Insulin Aspart 100 U/ml) With US and EU Insulin Aspart Comparator Products (NovoLog®/NovoRapid®) in Healthy Male Subjects
Brief Title: PK/PD Study of Gan & Lee Insulin Aspart Injection vs. US & EU NovoLog®/NovoRapid® in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GL-ASP-1008
Record Dates: First submitted 2020-01-15; First posted 2020-01-23 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes; Insulin; Diabetes Mellitus; Basal; Bolus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance | interventions — gallium nitrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Gan & Lee Insulin Aspart (Experimental): 100 units/mL, 3 ml prefilled pen
  Interventions: Drug: Gan & Lee Insulin Aspart
- NovoRapid® Insulin Aspart (Active Comparator): Product approved and marketed in the EU
  FlexPen100 units/mL prefilled pen
  Interventions: Drug: Gan & Lee Insulin Aspart
- NovoLog® Insulin Aspart (Active Comparator): Product approved and marketed in the US
  FlexPen100 units/mL prefilled pen
  Interventions: Drug: Gan & Lee Insulin Aspart

INTERVENTIONS:
Drug: Gan & Lee Insulin Aspart — All three IMPs will be administered as a 0.2 U/kg single dose subcutaneously in the periumbilical area.
  Other Names: NovoRapid® EU; NovoLog® US

SUMMARY:
Primary objective:

To demonstrate pharmacokinetic (PK) and pharmacodynamic (PD) equivalence of Gan & Lee Insulin Aspart Injection with both EU-approved NovoRapid® and US-licensed NovoLog® (Reference Products) in healthy male subjects

Secondary objectives:

To compare the PK and PD parameters of the three insulin aspart preparations

To evaluate the single dose safety and local tolerability of the three insulin aspart preparations

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent obtained before any trial-related activities. Trial-related activities are any procedures that would not have been done during normal management of the subject
2. Healthy male subjects
3. Age between 18 and 64 years, both inclusive
4. Body Mass Index (BMI) between 18.5 and 29.0 kg/m^2, both inclusive
5. Fasting plasma glucose concentration <= 5.50 mmol/L (100 mg/dL) at screening
6. Considered generally healthy upon completion of medical history, physical examination, vital signs, ECG and analysis of laboratory safety variables, as judged by the Investigator

Exclusion Criteria:

1. Known or suspected hypersensitivity to investigational medicinal products (IMPs) or related product
2. Previous participation in this trial. Participation is defined as randomized
3. Use of other investigational drugs within five half-lives for enrolment or receipt of any medicinal product in clinical development within 30 days before randomization in this trial, whichever is longer
4. History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.
5. Clinically significant abnormal values for haematology, biochemistry, coagulation, or urinalysis as judged by the Investigator
6. Increased risk of thrombosis, e.g subjects with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator
7. A positive result in the alcohol and/or urine drug screen at the screening visit
8. Positive to the screening test for Hepatitis Bs antigen or Hepatitis C antibodies and/or a positive result to the test for HIV-1/2 antibodies or HIV-1 antigen
9. Blood donation or blood loss of m ore than 500 mL within the last 3 months

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
AUCins.0-12h | 0 -12 hours
  PK endpoint: The area under the insulin concentration curve from 0 to 12 hours
Cins.max | 0 -12 hours
  PK endpoint: The maximum observed insulin concentration
AUCGIR.0-12h | 0 - 12 hours
  PD endpoint: The area under the glucose infusion rate curve from 0 to 12 hours
GIRmax | 0 - 12 hours
  PD endpoint: The maximum glucose infusion rate

SECONDARY OUTCOMES:
AUCins.0-2h | 0 - 2 hours
  PK endpoint: The area under the insulin concentration curve from 0 to 2 hours
AUCins.0-∞ | 0 - 12 hours
  PK endpoint: The area under the insulin concentration-time curve from 0 hours to infinity
tins.max | Up to Day 68
  PK endpoint: The time to maximum observed insulin concentration
t50%-ins(early) | Up to Day 68
  PK endpoint: The time to half-maximum insulin concentration before Cins.max
t50%-ins(late) | Up to Day 68
  PK endpoint: The time to half-maximum insulin concentration after Cins.max
t½ | Up to Day 68
  PK endpoint: The terminal serum elimination half-life calculated as t½=ln2/λz
λz | Up to Day 68
  PK endpoint: The terminal elimination rate constant of insulin
AUCGIR.0-2h | 0 - 2 hours
  PD endpoint: The area under the glucose infusion rate curve from 0 to 2 hours
tGIR.max | Up to Day 68
  PD endpoint: The time to maximum glucose infusion rate
tGIR.50%-early | Up to Day 68
  PD endpoint: The time to half-maximum glucose infusion rate before GIRmax
tGIR.50%-late | Up to Day 68
  PD endpoint: The time to half-maximum glucose infusion rate after GIRmax
PD endpoint | Up to Day 68
  time to onset of action
Safety and local tolerability | Up to Day 68
  Number of participants experiencing treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Matthew E Barton, PhD, Study Director — Gan & Lee Pharmaceuticals USA Corporation
Locations (1):
- Profil Mainz GmbH & Co. KG, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen W, Lu J, Plum-Morschel L, Andersen G, Zijlstra E, He A, Xie T, Li L, Hao C, Gan Z, Heise T. Pharmacokinetic and pharmacodynamic bioequivalence of Gan & Lee insulin analogues aspart (rapilin(R)), lispro (prandilin(R)) and glargine (basalin(R)) with EU- und US-sourced reference insulins. Diabetes Obes Metab. 2023 Dec;25(12):3817-3825. doi: 10.1111/dom.15281. Epub 2023 Sep 21. PMID 37735841